CLINICAL TRIAL: NCT04345861
Title: Randomized Trial Assessing Efficacy and Safety of Hydroxychloroquine Plus Azithromycin Versus Hydroxychloroquine for Hospitalized Adults With COVID-19 Pneumonia
Brief Title: Hydroxychloroquine Plus Azithromycin Versus Hydroxychloroquine for COVID-19 Pneumonia (COVIDOC Trial)
Acronym: COVIDOC
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: halted prematurely.
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RECHMPL20_168
Record Dates: First submitted 2020-04-05; First posted 2020-04-15 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: Coronavirus Infection; Pneumonia, Viral
Keywords: SARS-CoV2 virus; COVID-19; pneumonia; hydroxychloroquine; azithromycin
MeSH Terms: conditions — Coronavirus Infections; Pneumonia, Viral; COVID-19; Pneumonia | interventions — Hydroxychloroquine; Azithromycin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- monotherapy hydroxychloroquine (Active Comparator): Hydroxychloroquine 800mg (Day 1), 600mg (from Day 2 to Day 10) + placebo from Day 1 to Day 5
  Interventions: Drug: Hydroxychloroquine + placebo
- combination hydroxychloroquine + azithromycin (Experimental): Hydroxychloroquine 800mg (Day 1), 600mg (from Day 2 to Day 10) and azithromycin 500mg (Day 1 ), 250 mg (from day 2 to Day 5)
  Interventions: Drug: hydroxychloroquine + azithromycin

INTERVENTIONS:
Drug: Hydroxychloroquine + placebo — hydroxychloroquine : 800mg(Day1) then 600 mg (Day 2 to Day 11)
  Arms: monotherapy hydroxychloroquine
Drug: hydroxychloroquine + azithromycin — Combination hydroxychloroquine : 800mg(Day1) then 600 mg (Day 2 to Day 11) Azithromycin 500mg (day 1) then 250 mg (Day 2 to Day 5)
  Arms: combination hydroxychloroquine + azithromycin

SUMMARY:
Double blinded randomized clinical trial designed to evaluate the efficacy and safety of hydroxychloroquine combined with azithromycin compared to hydroxychloroquine monotherapy in patients hospitalized with confirmed COVID-19 pneumonia.

DETAILED DESCRIPTION:
The multi-centre COVIDOC study will evaluate the efficacy and safety of the use of hydroxychloroquine (10 days) combined with azithromycin (5 days) compared to hydroxychloroquine (10 days) in the the clinical evolution by the ordinal scale of 7 points in adults hospitalized outside Intensive care unit with pneumonia caused by infection by the SARS-CoV2 virus in France.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years old SARS CoV-2 Infection confirmed by positive virologic test realised in the 96 h before randomization
* Beginning of COVID-19 symptoms < 10 days at the time of randomization
* Presence of symptom(s) of COVID-19 : fever (température > or = 37,5°C) or respiratory sign(s) (cough, breathing discomfort) or recent anosmia
* Presence of TDM/radiographic signs or pneumonia
* Hospitalization out of ICU for COVID with: moderate clinical form (no oxygenotherapy) or non critical severe form (oxygenotherapy)

Exclusion Criteria:

* Absence of signed informed consent
* SpO2 < 90 % ambient air or < 94 % with oxygenotherapy > or = 3l/min
* Need of oxygenotherapy > 6 l/min or mechanical ventilation
* Need of hospitalization in ICU
* ALAT/ASAT > 5 LSN
* Renal failure (eGFR < 40 ml/min ) or dialysis
* Pregnancy or breastfeeding
* Retinopathy
* Known deficit in G6PD
* Cardiac rythm / lengthening QT disorders
* QT space lengthening on ECG with QTc > 450 ms
* Concomitant treatment :citalopram, escitalopram, hydroxyzine, domperidone, pipéraquine, anti-arhythmic class IA & III, antidepressive drugs,..

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2020-04-11 (Actual); Primary Completion 2021-02-09 (Actual); Study Completion 2021-04-09 (Actual)

PRIMARY OUTCOMES:
Time to clinical improvement of at least 1 level on the ordinal scale between Day 1 (day of the first administration of study drug) to Day 11 (day after last day of treatment). | up to Day 11
  Evaluation of the clinical status of patient defined by the Ordinal Scale of 7 points (score range from 1 to 7 , with 7 being the worst score)

SECONDARY OUTCOMES:
Clinical status assessed by ordinal scale | up to Day 29
  Evaluation of the clinical status of patient defined by the Ordinal Scale of 7 points at day 15 and day 29
transfer to ICU | up to Day 29
  Necessity for transfer to Intensive care unit
Length of hospital day | up to Day 29
  days from admission to hospital discharge
Hospital Mortality | Day 29
  incidence of all-cause mortality
Need to Mechanical Ventilation | up to Day 29
  Need to mechanical ventilation
Occurence of grade 3-4 adverse event | up to Day 29
  adverse reactions
QTc Lengthening | up to Day 11
  ECG
Evolution of pulmonary CT scan images | up to Day 11
  Thoracic CT scan : number and size of ground-glass opacifications on day 1 and day 11 Two independent pulmonary imagery experts will assess abnormalities according to a standardized framework

CONTACTS AND LOCATIONS:
Overall Officials: Jacques REYNES, MD,PhD, Principal Investigator — Montpellier University Hospital
Locations (1):
- Montpellier University hospital, Montpellier, France

IPD SHARING:
Plan to Share IPD: No